CLINICAL TRIAL: NCT01040429
Title: The Norwegian Study of Chronic Fatigue Syndrome in Adolescents: Pathophysiology and Intervention Trial
Acronym: NorCAPITAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Vegard Bruun Wyller, Associate professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NorCAPITAL.02
Record Dates: First submitted 2009-12-28; First posted 2009-12-29 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Fatigue Syndrome; Myalgic Encephalomyelitis
Keywords: Adolescent; Clonidine; Autonomic nervous system; Stress
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clonidine capsula (Active Comparator)
  Interventions: Drug: Clonidine
- Lactose capsula (Placebo Comparator)
  Interventions: Drug: Lactose capsula

INTERVENTIONS:
Drug: Clonidine — Day 1-56 (week 1-8): 25 microgram (1 capsula) x 2/day for patients < 35 kg; 50 microgram (2 capsula) x 2/day for patients > 35 kg.
  Day 57-63 (week 9): 25 microgram (1 capsula) x 1/day for patients < 35 kg; 25 microgram (2 capsula) x 2/day for patients > 35 kg.
  Arms: Clonidine capsula
Drug: Lactose capsula — Day 1-56 (week 1-8): 1 capsula x 2/day for patients < 35 kg; 2 capsula x 2/day for patients > 35 kg.
  Day 57-63 (week 9): 1 capsula x 1/day for patients < 35 kg; 1 capsula x 2/day for patients > 35 kg
  Arms: Lactose capsula

SUMMARY:
The purpose of this study IS to

* explore the underlying pathophysiology of chronic fatigue syndrome (CFS) in adolescents, particularly focusing on genetics, infections/immunology, endocrinology, autonomic control and cognitions
* to assess the effect of clonidine (a drug that attenuates sympathetic nervous activity) in adolescent CFS.

ELIGIBILITY:
Inclusion Criteria:

* Persisting or constantly relapsing fatigue lasting 3 months or more.
* Functional disability resulting from fatigue to a degree that prevent normal school attendance

Exclusion Criteria:

* Another disease process or current demanding life event that might explain the fatigue
* Another chronic disease (in particular pheochromocytoma, polyneuropathy, Renal insufficiency)
* Permanent use of pharmaceuticals (including hormone drugs)
* Permanently bed-ridden
* Positive pregnancy test
* Evidence of reduced cerebral and/or peripheral circulation due to vessel disease
* Know hypersensitivity towards clonidine or inert substances (lactose, sakkarose) in capsula
* Abnormal ECG (in particular bradyarrythmias due to sick sinus syndrome or AV-block. Isolated ectopic beats do not lead to exclusion)
* Supine heart rate < 50 beats/min
* Supine systolic blood pressure < 85 mmHg
* Systolic blood pressure fall upon standing > 30 mmHg

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2010-02; Primary Completion 2012-06 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Mean steps/day count during one week | 8 weeks after inclusion

SECONDARY OUTCOMES:
Fatigue scores | 8 and 30 weeks after inclusion
Pain scores | 8 and 30 weeks after inclusion
Algometer testing response | 8 and 30 weeks after inclusion
Autonomic symptom scores | 8 and 30 weeks after inclusion
Quality of life-score | 8 and 30 weeks after inclusion
Disability scores | 8 and 30 weeks after inclusion
School attendance | 8 and 30 weeks after inclusion
Mean steps/day count during one week | 30 weeks after inclusion
Scores on cognitive function tests | 8 and 30 weeks after inclusion
The change in mean arterial pressure (MAP) during head-up tilt-test | 8 and 30 weeks after inclusion
The change in heart rate during head-up tilt-test | 8 and 30 weeks after inclusion
The change in LF/HF-ratio (a measure of autonomic control) during head-up tilt-test | 8 and 30 weeks after inclusion
Hormonal levels (inluding tryptophan metabolites) | 8 and 30 weeks after inclusion
Microbiological analyses | 8 and 30 weeks after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Bruun Wyller, MD, PhD, Principal Investigator — Dept. of Pediatrics, Oslo University Hospital, Norway
Locations (1):
- Dept. of Pediatrics, Oslo University Hospital Rikshospitalet, Oslo, Oslo County, Norway

REFERENCES:
- [Background] Wyller VB, Eriksen HR, Malterud K. Can sustained arousal explain the Chronic Fatigue Syndrome? Behav Brain Funct. 2009 Feb 23;5:10. doi: 10.1186/1744-9081-5-10. PMID 19236717
- [Background] Wyller VB, Due R, Saul JP, Amlie JP, Thaulow E. Usefulness of an abnormal cardiovascular response during low-grade head-up tilt-test for discriminating adolescents with chronic fatigue from healthy controls. Am J Cardiol. 2007 Apr 1;99(7):997-1001. doi: 10.1016/j.amjcard.2006.10.067. Epub 2007 Feb 16. PMID 17398200
- [Derived] Asprusten TT, Sletner L, Wyller VBB. Are there subgroups of chronic fatigue syndrome? An exploratory cluster analysis of biological markers. J Transl Med. 2021 Jan 30;19(1):48. doi: 10.1186/s12967-021-02713-9. PMID 33516248
- [Derived] Wyller VB, Nguyen CB, Ludviksen JA, Mollnes TE. Transforming growth factor beta (TGF-beta) in adolescent chronic fatigue syndrome. J Transl Med. 2017 Dec 4;15(1):245. doi: 10.1186/s12967-017-1350-1. PMID 29202780
- [Derived] Nguyen CB, Alsoe L, Lindvall JM, Sulheim D, Fagermoen E, Winger A, Kaarbo M, Nilsen H, Wyller VB. Whole blood gene expression in adolescent chronic fatigue syndrome: an exploratory cross-sectional study suggesting altered B cell differentiation and survival. J Transl Med. 2017 May 11;15(1):102. doi: 10.1186/s12967-017-1201-0. PMID 28494812
- [Derived] Wyller VB, Vitelli V, Sulheim D, Fagermoen E, Winger A, Godang K, Bollerslev J. Altered neuroendocrine control and association to clinical symptoms in adolescent chronic fatigue syndrome: a cross-sectional study. J Transl Med. 2016 May 5;14(1):121. doi: 10.1186/s12967-016-0873-1. PMID 27149955
- [Derived] Fagermoen E, Sulheim D, Winger A, Andersen AM, Gjerstad J, Godang K, Rowe PC, Saul JP, Skovlund E, Wyller VB. Effects of low-dose clonidine on cardiovascular and autonomic variables in adolescents with chronic fatigue: a randomized controlled trial. BMC Pediatr. 2015 Sep 10;15:117. doi: 10.1186/s12887-015-0428-2. PMID 26357864
- [Derived] Winger A, Kvarstein G, Wyller VB, Sulheim D, Fagermoen E, Smastuen MC, Helseth S. Pain and pressure pain thresholds in adolescents with chronic fatigue syndrome and healthy controls: a cross-sectional study. BMJ Open. 2014 Oct 6;4(9):e005920. doi: 10.1136/bmjopen-2014-005920. PMID 25287104
- [Derived] Sulheim D, Fagermoen E, Winger A, Andersen AM, Godang K, Muller F, Rowe PC, Saul JP, Skovlund E, Oie MG, Wyller VB. Disease mechanisms and clonidine treatment in adolescent chronic fatigue syndrome: a combined cross-sectional and randomized clinical trial. JAMA Pediatr. 2014 Apr;168(4):351-60. doi: 10.1001/jamapediatrics.2013.4647. PMID 24493300
- [Derived] Fagermoen E, Sulheim D, Winger A, Andersen AM, Vethe NT, Saul JP, Thaulow E, Wyller VB. Clonidine in the treatment of adolescent chronic fatigue syndrome: a pilot study for the NorCAPITAL trial. BMC Res Notes. 2012 Aug 7;5:418. doi: 10.1186/1756-0500-5-418. PMID 22871021